CLINICAL TRIAL: NCT01655498
Title: A Clinical Evaluation of the LivSure Vaginal Bowel Control (VBC) System for the Treatment of Fecal Incontinence in Women.
Brief Title: A Clinical Evaluation of a Vaginal Bowel Control System for the Treatment of Fecal Incontinence in Women (LIFE)
Acronym: LIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pelvalon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA003
Record Dates: First submitted 2012-07-24; First posted 2012-08-02 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence; bowel control
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaginal Bowel Control (Experimental): A vaginal bowel control system intended to manage fecal incontinence.
  Interventions: Device: vaginal bowel control system (LivSure)

INTERVENTIONS:
Device: vaginal bowel control system (LivSure)
  Other Names: LivSure System; Eclipse™ System

SUMMARY:
The objective of this study is to obtain preliminary efficacy and safety data on the use of the LivSure System (now called the "Eclipse™ System") in women with fecal incontinence.

ELIGIBILITY:
Inclusion Criteria:

* History of FI for at least 6 months
* Baseline diary requirement for min # of FI episodes in a two-week period
* Ability to manage investigational device insertion and removal
* Successful fitting of study device
* Willing and able to give written informed consent to participate in the study

Exclusion Criteria:

* Chronic rectal, anal or pelvic pain
* Any vaginal prolapse that extends beyond the plane of the hymen.
* Previous rectal or pelvic floor surgery within the last 12 months (24 months in the case of cancer)
* Congenital anorectal malformation
* Chronic watery diarrhea unmanageable by drugs or diet as primary cause of FI
* Inflammatory bowel disease
* Presence of a vaginal, anal, rectal or urethral fistula or anastomosis
* Presence of a vaginal, rectal or bladder tumor
* Presence of an open wound or tear in the vagina or anus by exam
* Presence or history of rectovaginal fistula
* Atrophic vaginal tissue as determined by symptoms or visualization
* Current vaginal or urinary infection requiring treatment
* History of recurrent urinary or vaginal infections
* Subject is currently pregnant or planning pregnancy in next 5 months
* Concurrent use of any intra-vaginal device that would interfere with LivSure (now called Eclipse) placement or wearing
* Any significant medical condition (e.g., significant psychiatric or neurological disorders, active alcohol/drug abuse, etc.) or other factor that the investigator believes would interfere with study participation and/or increase subject risk

Ages: 19 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-08; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Richter, PhD, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Matthews CA, Varma MG, Takase-Sanchez MM, Hale DS, Van Drie D, Muir T, Wells E, Jannelli M, Richter HE. Characteristics Associated With Successful Fitting of a Vaginal Bowel Control System for Fecal Incontinence. Female Pelvic Med Reconstr Surg. 2016 Sep-Oct;22(5):359-63. doi: 10.1097/SPV.0000000000000290. PMID 27564386
- [Derived] Richter HE, Matthews CA, Muir T, Takase-Sanchez MM, Hale DS, Van Drie D, Varma MG. A vaginal bowel-control system for the treatment of fecal incontinence. Obstet Gynecol. 2015 Mar;125(3):540-547. doi: 10.1097/AOG.0000000000000639. PMID 25730213

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited primarily through Investigators' private practices with some additional participants recruited through IRB approved advertisements between 14 Aug 2012 through Nov. 2013.
Pre-assignment Details: 200 subjects were consented:
  Pre-fitting screen fails: vaginal anatomical exclusions (13), logistics issues (12), LTFU (5), other (16).
  Baseline diary screen fails: (44).
  Post-fitting screen fails: unsatisfactory fit (28), unable to manage device (4), LTFU (1), logistics issues (2), withdrawal (14).
Groups:
- All Subjects: All subjects who completed the fitting process and entered the treatment period, comprised the Intent-to-treat population.
Period: Overall Study
Arm/Group | All Subjects
Started | 61
Completed | 56
Not Completed | 5
Not completed — Unrelated health issue | 2
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All subjects who were successfully fit with the VBC device (now called Eclipse)
Groups:
- All Subjects: All subjects who completed the fitting process (a screening criteria) and entered the treatment period.
Arm/Group | All Subjects
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 45
  Asian | 2
  Black | 10
  American Indian or Alaska Native | 0
  Hispanic or Latino | 3
  Natrive Hawaiian or Other Pacific Islander | 0
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 61
Body Mass Index [Number; unit: participants]
  <18.5 | 2
  18.5-24.9 | 20
  25.0-29.9 | 21
  >29.9 | 18
Previous Gynecologic Surgeries [Number; unit: participants]
  Hysterectomy | 29
  Prolapse surgery | 5
  Urinary incontinence surgery | 9
  Other gynecologic surgery | 25
Sexual Activity [Number; unit: participants]
  Greater than or equal to 1 x month | 27
  Less than 1 x per month | 33
  Not reported | 1
Parity [Median (Full Range); unit: events]
  No. of pregnancies | 2 [0 to 12]
  No. of vaginal births | 2 [0 to 4]
Menopause Status [Number; unit: participants]
  Pre-menopause | 7
  Peri-menopause | 2
  Post-menopause | 51
  Not reported | 1
Number of FI episodes in 2-week period [Mean (Standard Deviation); unit: episodes] | 11.7 (9.1)
FI Symptom Duration [Number; unit: participants]
  6 months - 5 years | 35
  > 5 years | 26
Previous treatment for FI [Number; unit: participants]
  Surgery | 4
  Surgical implant of electrical stimulator [n=60] | 1
  Biofeedback | 11
  Other [n=60] | 6

OUTCOME MEASURES:

1. Primary Outcome: Frequency of FI Episodes
Description: Subjects with at least a 50% reduction in FI episodes (major or minor soiling)
Time Frame: 1 Month
Population: Subjects who were successfully fit with the VBC device.
Measure: Number; unit: percentage of participants
Groups:
- Subjects Fit With the VBC Device [ITT]: ITT cohort is defined as all subjects who were successfully fit with a VBC device (now called Eclipse Insert) during the Fitting Period
- Subject Fit With the VBC Device [PP]: Per Protocol cohort is defined all all subjects who were successfully fit with a VBC device (now called Eclipse Insert) during the Fitting Period who also completed the study without any major protocol deviations
Arm/Group | Subjects Fit With the VBC Device [ITT] | Subject Fit With the VBC Device [PP]
Number analyzed (Participants) | 61 | 56
percentage of participants | 79 | 86

2. Secondary Outcome: Number of Incontinent Days
Description: Change in number of incontinent days while wearing the device during the 2-week assessment period as compared to the baseline 2-week assessment period
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subject Fit With the VBC Device [PP]
Number analyzed (Participants) | 56
days
  # Episodes reported at 1 Month | 2.1 (2.9)
  # Episodes reported at Baseline | 11.6 (9.5)

3. Secondary Outcome: Device-related Adverse Events
Description: The number of overall adverse events rated as probably or definitely related to the study device.
Time Frame: 1month
Population: All subjects who were exposed to the VBC device (now called Eclipse) during the Treatment Period.
Measure: Number; unit: events
Groups:
- ITT Cohort [N=61]: All subjects who entered the Treatment Period.
Arm/Group | ITT Cohort [N=61]
Number analyzed (Participants) | 61
events | 18

ADVERSE EVENTS:
Time Frame: 1 month Treatment Period
Groups:
- ITT Cohort [N=61]: Adverse Events reported during the Screening and 1-Month Treatment Period.
Arm/Group | ITT Cohort [N=61]
Serious Adverse Events (participants affected / at risk) | 1/61
Other Adverse Events (participants affected / at risk) | 36/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ITT Cohort [N=61] (N=61)
Flu symptoms (Infections and infestations) | 1 — Required hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITT Cohort [N=61] (N=61)
Pelvic cramping or discomfort (Reproductive system and breast disorders) | 16 (16)
Pelvic pain (Reproductive system and breast disorders) | 6 (6)
Urinary incontinence (Renal and urinary disorders) | 6 (6)
Difficulty with Stool Evacuation (Gastrointestinal disorders) | 4 (4)
Urinary urgency or frequency (Renal and urinary disorders) | 4 (4)
Vaginal Spotting (Reproductive system and breast disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days